CLINICAL TRIAL: NCT02885402
Title: Functional Exploration of Cartilage in Patients With Osteoarthritis of the Knee Through MRI Sodium ( 23Na )
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-05; 2016-A00427-44 (Other: Ansm)
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteoarthritis patient (Experimental)
  Interventions: Other: MRI Sodium ( 23Na )
- Healthy volunteers (Placebo Comparator)
  Interventions: Other: MRI Sodium ( 23Na )

INTERVENTIONS:
Other: MRI Sodium ( 23Na )

SUMMARY:
Osteoarthritis is a degenerative disease of hyaline cartilage not associated with an infection or an inflammatory process that affects millions of people. The first symptoms usually appear from 40-50 years and at this point, conventional radiological tests provide diagnostic elements relatively late, poorly correlated with pain relief and providing no functional information. In this context, there is a real need for imaging techniques for early detection of osteoarthritic changes in a still reversible stage for faster support and MRI appears to be the tool of choice.

Conventional proton MRI sequences already allow improved detection possibilities compared to conventional radiology and CT arthrography supplanted. They nevertheless remain insufficient to identify incipient lesions or paradoxically to the point of too advanced lesions. Due to recent technological advances, exploration MRI other nuclei such as sodium is now possible. Quantitation of sodium in the cartilage by sodium MRI allow quantifying proteoglycan loss and ultimately a gradation osteoarthritic reached.

This project's main objective is to quantify the biochemical changes (sodium content) occurring at different stages of osteoarthritis defined by clinical algofunctional scores (Lequesne) and conventional radiographic scores (Kellgren and Lawrence).

ELIGIBILITY:
Inclusion Criteria:

* Patient with osteoarthritis

Exclusion Criteria:

* patient with contraindication for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of sodium released in osteoarthritis patient vs healthy volunteers | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre MATTEI, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille; Urielle Desalbres, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No